CLINICAL TRIAL: NCT07275983
Title: Total Knee Replacement Under Spinal Anesthesia, Comparison of Postoperative Recovery Versus General Anesthesia: A Retrospective Single-Center Observational Comparative Superiority Study
Brief Title: Total Knee Replacement Under Spinal Anesthesia, Comparison of Postoperative Recovery Versus General Anesthesia
Acronym: PTG-RachiVsAG
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9305
Record Dates: First submitted 2025-03-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Total Knee Replacement
Keywords: knee; Total Knee Replacement; Spinal Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intraoperative anesthetic management for total knee replacement (TKR) can be performed under general or spinal anesthesia. These two techniques have their own characteristics and may impact postoperative recovery differently. However, there are no studies in the literature analyzing postoperative functional recovery after TKR surgery according to the type of anesthesia. The objective of this study is to compare postoperative recovery, assessed by the QoR-15F score, in patients undergoing TKR under spinal anesthesia versus surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older (no upper age limit)
* Underwent total knee replacement surgery between January 1, 2020 and June 30, 2023
* Assessed using the QoR-15F score

Exclusion Criteria:

* Subject (and/or their legal representative, if applicable) who expressed their opposition to the reuse of their data for scientific research purposes.
* Revision, emergency, oncological, bilateral, or septic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject having total knee replacement surgery between January 1, 2020 and June 30, 2023
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
QoR-15F score | at Day 1, Day3, Day 14, and Day 28 postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésiologie - Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France